CLINICAL TRIAL: NCT05731960
Title: A Randomized Controlled Trial Evaluating the Effect of Intravenous Dexamethasone on the Duration of Spinal Anesthesia as Part of a Multimodal Antiemetic Strategy for Enhanced Recovery After Cesarean Delivery
Brief Title: Evaluating the Effect of Intravenous Dexamethasone on the Duration of Spinal Anesthesia After Cesarean Delivery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: IWK Health Centre (Other)
Responsible Party: Principal Investigator, Allana, Principal Investigator, IWK Health Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1028461
Record Dates: First submitted 2023-01-17; First posted 2023-02-16 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Spinal Anesthesia; Dexamethasone
Keywords: spinal anesthesia; dexamethasone; motor block
MeSH Terms: interventions — Dexamethasone; Metoclopramide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexamethasone (Group SD) (Experimental): 10 mg IV dexamethasone x1
  Interventions: Drug: Dexamethasone
- Metoclopramide (Group SM) (Active Comparator): 10 mg IV metoclopramide x1
  Interventions: Drug: Metoclopramide

INTERVENTIONS:
Drug: Dexamethasone — 10 mg IV dexamethasone provided immediately after spinal anesthesia
  Arms: Dexamethasone (Group SD)
Drug: Metoclopramide — 10 mg IV metoclopramide provided immediately after spinal anesthesia
  Arms: Metoclopramide (Group SM)

SUMMARY:
The goal of this clinical trial is to determine the effects of intravenous (IV) dexamethasone on spinal anesthesia in healthy women having an elective Cesarean delivery (CD) at the IWK Health Centre. The main questions it aims to answer are:

1. What effect does IV dexamethasone have on the resolution of motor blockade in patients having spinal anesthesia for elective CDs?
2. What effect does IV dexamethasone have on the sensory recovery of spinal blockade, the total hydromorphone requirement in the first 24 h postoperatively, the incidence of pruritis perioperatively, and the incidence of nausea and vomiting?

The spinal anesthesia technique will be standardized and will be administered as per routine care at IWK Health. Computer generation will randomize patients to either Group SD, who will receive IV dexamethasone, or group SM who will receive IV metoclopramide, an alternative anti-emetic, immediately after spinal anesthesia by the attending anesthesia provider. Each patient will receive ondansetron, a second anti- emetic as recommended for Enhanced Recovery After Surgery (ERAS) protocol. Participant sensation, pain, nausea, pruritus, and motor blockade will be assessed in recovery. The patient's sensation and Bromage score will be assessed every 15 minutes until sensation is reached at L3 and a Bromage score of 4 is achieved.

The investigators will determine if there is a difference between groups regarding motor blockade, the length of time of spinal anesthesia, and side effects after CD.

DETAILED DESCRIPTION:
Background:

Enhanced Recovery After Surgery (ERAS) is a concept that aims to achieve faster patient recovery and fewer complications after major surgery. Spinal anesthesia is a technique widely used for Cesarean Delivery (CD), where a local anesthetic is administered along with opioids such as fentanyl and morphine. Antiemetic agents have been used prophylactically during CD under spinal anesthesia. The efficacy of combination antiemetic agents to prevent nausea and vomiting in patients who underwent CD has been established, hence, a multi-modal anti-emetic approach has been advocated for ERAS for CD.

Dexamethasone is a corticosteroid that has been found to significantly prevent nausea and vomiting and decrease postoperative pain. Dexamethasone has been shown to prolong the durations of sensory and motor blockade for peripheral nerve blocks. Despite the knowledge that dexamethasone is a useful adjunct for extending local anesthetic duration and reducing postoperative pain, only one study has examined its application in spinal anesthesia for CD. In this study, authors found 8mg of IV dexamethasone increased the mean duration of sensory block by 56 minutes, which was highly significant. The extended duration of anesthesia can have several unintended consequences such as extending stay in the post anesthesia recovery unit (PACU), impairing mother and baby bonding, and utilizing healthcare resources as nurses have to stay with the patient longer limiting the ability to complete another elective CD.

Recognizing the perioperative movement towards adopting ERAS strategies, dexamethasone will be a routine adjunct to prevent spinal associated nausea and vomiting. Formally quantifying the effect IV dexamethasone has on spinal anesthesia for CD will help anesthesia providers decide whether to administer IV dexamethasone intraoperatively. For example, if providers are hoping to extend the length of the spinal blockade (prolonged surgical duration) they could choose dexamethasone as the second multi-modal antiemetic. Alternatively, anesthesia providers could omit IV dexamethasone, and use an alternative anti- emetic such as metoclopramide, to promote rapid discharge from the PACU, improving perioperative efficiency and health utilization.

The investigators hypothesize that in healthy parturients having elective CD, 10 mg IV dexamethasone will increase the duration of motor blockade from spinal anesthesia using 0.75% bupivacaine, lengthening the time spent in PACU.

Design & Procedure:

This is a randomized double-blind controlled clinical trial in non-laboring parturients presenting for elective CD.

The spinal anesthesia technique will be standardized and will be administered as per routine care at IWK Health. Each patient will receive 12 mg of 0.75% hyperbaric bupivacaine with 10 micrograms of fentanyl and 100 micrograms of epidural morphine via a 25-gauge Whitacre spinal needle. Computer generation will randomize patients to either Group SD, who will receive IV dexamethasone 10 mg (1mL), or group SM who will receive IV metoclopramide 10 mg (2 mL) (alternative anti-emetic), immediately after spinal anesthesia by the attending anesthesia provider. Additionally, each patient will receive ondansetron 4mg IV, immediately after spinal anesthesia (second anti-emetic as recommended for ERAS protocol). If a third anti-emetic is required for ongoing nausea and vomiting in the operating room or PACU, dimenhydrinate 12.5- 25 mg IV can be provided for both groups. If a fourth anti-emetic is required for ongoing nausea and vomiting in the operating room or PACU, haloperidol 0.5mg IV can be provided for both groups. All anti-nausea medications administered will be tracked on the data collection record (DCR).

The randomization assignments will be placed in a sealed envelope by a research staff member who is not participating in clinical data collection. The randomization log will be kept in a secure/locked research office. The randomization envelope will be provided to the attending anesthesiologist by a research team member on the morning of surgery. All drugs will be prepared and administered by the attending anesthesiologist, who will not be blind. The patient and research team assessor will be blinded to treatment allocation.

Sensation will be tested using ice and quality of motor block will be assessed using modified Bromage score. In PACU, research personnel, unaware of the subject's randomization, will assess motor blockade unilaterally every 15 minutes until a Bromage score of 3 is present. That time will be entered on the DCR, and the patient will be assessed more frequently (every 3-5 minutes) until a Bromage of 4 is achieved and confirmed bilaterally with a second assessment 1-minute later. If needed, assessments will continue to occur every 3-5 minutes until a Bromage score of 4 is reached bilaterally. Sensation will be assessed every 15 minutes unilaterally. When sensation is reached at L3, a bilateral assessment will be taken, and the time will be recorded. If needed, assessments will continue to occur every 15 minutes. The time will be recorded on the DCR when sensation at L3 is reached bilaterally.

Numeric Rating Scale (NRS) scores for pain and nausea intensity will be collected every hour postoperatively until a Bromage score of 4 is achieved. The time of opioid use and total opioid dose in the first 24 h will be recorded during the PACU stay and from medical chart review. The incidence of pruritus (itching) and vomiting will also be assessed prior to PACU discharge.

Data Analysis:

In keeping with CONSORT guidelines, all subjects enrolled will be included in an intention to treat analysis. Descriptive statistics will be expressed as mean +/- standard deviation. Demographics (height, weight, etc.) will be analyzed using Student's t-test. Nonparametric testing (Mann-Whitney U test) will be used to evaluate NRS pain scores, opioid consumption and sensory and motor duration. Categorical data (nausea and vomiting) will be analyzed using the x2 test or Fisher's exact test, as appropriate. The investigators will perform the statistical analysis with the assistance of the consulting departmental statistician.

With power of 90% and confidence interval of 95% (α = 0.05), a clinically meaningful change in recovery time of 15 minutes with a (generous) anticipated standard deviation of 33, 116 participants are required (58 per group). It is anticipated that the standard deviation could be smaller than this, which would mean that the investigators could be powered to detect a 15-minute difference at α = 0.05 with fewer than 116 participants. 116 is a conservative estimate to ensure that the investigators have the power needed to test the primary hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Non-emergent Caesarean Delivery with planned spinal anesthesia
* American Society of Anesthesia physical status class < III
* Age ≥18 years
* Term gestational age (≥37weeks)
* Singleton pregnancy
* Moderate English language fluency

Exclusion Criteria:

* Obesity (BMI ≥ 45kg/m2)
* Height < 5'0"
* Patients with significant obstetric or neonatal co-morbidities (i.e., severe maternal cardiac disease, preeclampsia, fetal anomalies)
* Opioid tolerance or sensitivity
* Intolerance to non-steroidal anti-inflammatory drugs (NSAIDs)
* Contraindication to neuraxial analgesia (i.e., coagulopathy, infection, neuropathy)
* Abnormal spinal anatomy (i.e., severe scoliosis, spina bifida, spinal instrumentation)
* Use of chronic steroids
* A physical or psychiatric condition which impairs cooperation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant
Enrollment: 192 (Estimated)
Dates: Start 2023-03-06 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Resolution of motor blockade assessed by the Bromage motor blockade score | Upon entrance to PACU until a Bromage score of 4 is achieved bilaterally
  A Bromage score is quantified from 1 to 4, where a score of 1 indicates a complete block and patients are unable to move their feet or knees. A score of 2 indicates patients are able to only move their feet, while a score of 3 indicates slight knee movement and movement of the feet. A score of 4 indicates full flexion of the knees and feet. When a Bromage score of 3 is reached, assessments will instead occur every 3-5 minutes until a Bromage of 4 is achieved and confirmed bilaterally with a second assessment 1-minute later. If needed, assessments will continue to occur every 3-5 minutes until a Bromage score of 4 is reached bilaterally. The time will be recorded to specify the hour and minute of each assessment. A Bromage score of 4 indicates the endpoint.

SECONDARY OUTCOMES:
Sensory recovery of spinal blockade assessed by dermatome testing | Upon entrance to PACU until sensory is achieved bilaterally at L3
  Dermatome assessments using ice will occur every 15-minutes unilaterally. When sensation is reached at L3 (the greater trochanter region of the femur), a bilateral assessment will be taken, and the time will be recorded. If needed, assessments will continue to occur until sensation has been reached at L3 bilaterally. The time will be recorded to specify the hour and minute of each assessment.
Total opioid requirement (mg) in the first 24 hours postoperatively | Retrieved at 24 hours following spinal anesthesia.
  Recorded from the Intraoperative Anesthesia Information Management System (in milligrams, mg).
Pain scores assessed by NRS | Every hour postoperatively until a Bromage score of 4 is achieved.
  Numeric Rating Scale (NRS) is quantified as 0-10, where 0 is none, 1-3 is mild, 4-6 is moderate, and 7-10 is severe, where 10 represents the worst pain imaginable.
Nausea intensity scores assessed by NRS | Every hour postoperatively until a Bromage score of 4 is achieved.
  Numeric Rating Scale (NRS) is quantified as 0-10, where 0 is none, 1-3 is mild, 4-6 is moderate, and 7-10 is severe, where 10 represents the worst nausea intensity imaginable.
Incidence of pruritis (itching) | Post-operatively at time of PACU discharge
  Assessed by asking participants "yes" or "no"
Incidence of vomiting | Post-operatively at time of PACU discharge
  Assessed by asking participants "yes" or "no"

CONTACTS AND LOCATIONS:
Overall Officials: Allana Munro, MD FRCPC, Principal Investigator — IWK Health; Kwesi Kwofie, MD FRCPC, Principal Investigator — IWK Health
Locations (1):
- IWK Health Centre, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No